CLINICAL TRIAL: NCT04668560
Title: Improving Wellbeing, Health and Work Adherence Effects of the 5 Ways to Wellbeing Course
Brief Title: Effects of the 5 Ways to Wellbeing Course Effects of the 5 Ways to Wellbeing Course
Acronym: FiveWays
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: The Dam Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 59001
Record Dates: First submitted 2020-12-02; First posted 2020-12-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Wellbeing; Quality of Life; Mental Health Wellness 1

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Masking Description: Behavioural intervention, masking N/A
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Course intervention, six weeks wellbeing course
  Interventions: Behavioral: Five ways to wellbeing course
- Control (No Intervention): Follow-up as usual

INTERVENTIONS:
Behavioral: Five ways to wellbeing course — A behavioural course over six sessions. Teaching the participants in doing avtivities to promote wellbeing
  Arms: Intervention

SUMMARY:
Norway and other Western industrialized countries are facing major challenges in terms of preventable health problems, high work absence, largescale demographic changes and rising social inequalities in health. This project addresses the need for effective means to meet these important challenges. The project will scientifically evaluate The 5 Ways to Wellbeing course (5Ways), a novel measure aiming to promote wellbeing and integration, health and work adherence. Subjective wellbeing is systematically and prospectively related to important individual and societal outcomes, including social connectedness and integration, innovation, productivity, work performance, healthy behaviours, health and longevity. Promotion of wellbeing may therefore contribute to address the urgent societal ailments of today. Intervention effects and cost effectiveness of the 5Ways will be examined in-depth in four real-life settings, using quantitative methods. Specifically, we will investigate course impact wellbeing, health and work adherence among users of The Norwegian Labour and Welfare Administration (NAV) and clients in Healthy Life Centres. If effective, the course may be implemented nationwide and contribute to increase wellbeing and work participation. Findings from the study may thus contribute to enable municipalities and workplaces to make better priorities for promoting work presence, reducing suffering and improving mastery and quality of life among their inhabitants.

DETAILED DESCRIPTION:
Sample:

The sample consists of individuals attending the 5Ways course offered in Healthy Life Centres HLCs (N=500) and in NAV centres (N=100), and two groups of control subjects. The control groups include i) 1200 individuals participating in the FLS study and ii) 100 individuals in NAV receiving follow up as usual. The target group for the 5Ways course consists of individuals with, or at high risk of disease, who need support in health behaviour change and in coping with health problems and chronic disease. HLCs are interdisciplinary primary health care services that offer effective measures for people who need support in health behaviour change and in coping with health problems and chronic disease. All 5Ways course participants in HLCs will be invited to enrol in the study. In total, the investigators assume that altogether 500 participants from HLCs will be included in the study. The second group of course participants will include individuals on sick leave, work assessment allowance and disability pension who receive the 5Ways course through NAV. NAV currently administers a third of the national budget through schemes such as unemployment benefit, work assessment allowance, pensions, etc. The NAV participants will be randomised into an intervention group or a control group. Exclusion criteria for participation in the course include impaired cognitive functioning and severe mental illness.

The Course Intervention. The participants will attend the course for 2.5 hours across six weeks, one session dedicated to each of the five actions, and the last session for summarising, sharing and evaluating. The course is ready to be implemented. The course leaders are HLC coaches and NAV employees, with a minimum of three years of relevant education who are certified to run the 5Ways course. Course leader training consists of a two-day intensive, highly standardized training program. All course leaders receive a comprehensive manual to be followed through the course. The participants receive standardised course material.

The Pilot Study. During spring 2018, a pilot study was conducted on the 5Ways course in 12 HLCs in the South-Eastern part of Norway. A total of 89 participants completed the evaluation questionnaire. The evaluation report concluded that the participants were highly satisfied (score: 8.7/10), intended to continue to practice what they had learnt and experienced improved wellbeing.

Research hypotheses.

The investigators hypothesize that participating in the 5Ways course will improve wellbeing, physical and mental health, mastery and social participation, and thus ultimately reduce the burden of disease, reduce utilisation of health care services, and increase work participation. The investigators will examine effects on all outcome measures in different vulnerable groups short term, after completion of the course, and long term, after 6 and 15 months, on participants in HLCs and users on welfare benefits in the NAV system. The investigators have three main hypotheses:

1. The 5Ways course improves wellbeing, physical and mental health and mastery, short term and long term.
2. The 5Ways course reduces loneliness, strengthens social integration, and increases social support, short term and long term.
3. The 5Ways course increases return to work and long-term work participation in individuals on sick leave or welfare benefits.

Design. The design is a prospective controlled comparative study, using two different groups, with and without randomisation. Group 1: Participants referred to HLCs, and group 2: Individuals receiving welfare benefits from The Norwegian Labour and Welfare Administration (NAV). The long-term results from group 1 will be compared to a group of HLC users not offered the course (i.e., participating in the ongoing FLS-study).

A randomised controlled trial (RCT) was originally planned for both HLCs and NAV. However, both end users and HLC coaches urged the investigators to avoid randomisation in HLCs. HLC participants often need to build up the courage to seek help over time. Randomisation to no/delayed course (e.g., waiting list control) was therefore considered unethical. In NAV, the users have not requested health care services. Hence, not being offered the course is "treatment as usual". By conducting a study in NAV, the project meets the gold standard of using a RCT.

Group 1. Participants referred to HLCs, receiving regular HLC services, will be offered the course and invited to participate in the study. The HLC coaches will be responsible for the recruitment of course participants. Control for group 1. A large-scale study on effects of participation in HLCs, the FLS-study (Frisklivsstudien, N=1200) is about to be completed. The FLS participants are similar to our group 1 in terms of characteristics. The FLS study also include some of the outcome measures to be used in our planned study. The FLS data thus give the investigators the opportunity to compare the 5Ways course with effects of basic HLC interventions (i.e., 12 weeks follow-up of health behaviour change by a HLC coach). Group 2. People on welfare benefits, such as long-term sick leave and disability pensions, in the NAV-system will be recruited by NAV employees and randomised into two groups, an intervention group and a control group. The intervention group will participate in the course, and the control group will be followed up as usual in NAV (i.e., not offered the course). In groups 1 and 2 the participants will receive the questionnaire at the start of the course, at the end of the course, at 6 months and at 15 months. Four measurement waves enable the investigators to model long-term changes in the outcome variables after the intervention using multilevel methods, as this requires at least three measurements in the follow up phase. Although one would expect some dropout, all the available data will be useful in this approach, as it does not require listwise deletion of individuals with missing data. There will be approximately 70 courses altogether, 60 in HLCs and 10 in NAV. This will allow the investigators to investigate the extent to which course effects and the subsequent developmental trajectories in participants differ between groups. The investigators can also account for this variability by including level two predictors, such as the course leaders' fidelity to the manual. Follow-up data collected after 15 months will be compared to the 15 months' follow-up data in the FLS study. This design enables the investigators to examine potential effects in two ways: 1. Examine the added effect of the 5Ways course to ordinary HLC services at 15 months. 2. Examine the effect of the course in a group of individuals on welfare benefits compared to a control group in NAV.

Instruments. Subjective wellbeing is the primary outcome in this study. Secondary outcome measures are physical and mental health, mastery, social integration, physical activity, use of health care services and work adherence. Measurement tools in the recent report on recommendations for a better quality of life measurement system, will be used. These include OECD's recommended minimum-tool for assessing quality of life, Diener's flourishing scale, Satisfaction With Life Scale (SWLS), Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS), Pearlin and Schoolers Mastery Scale, Patient Health Questionnaire (PHQ-2), Oslo Social Support Scale (OSS-3) and Hopkins Symptom Checklist (HSCL). In addition, the investigators will use The Short Form Survey-12 (SF-12) and standardised questions on physical activity from the North-Trøndelag Health Survey (HUNT). The latter questions are used in the FLS-study. Background data such as age, gender, education, work attachment, economy and relationship status will also be collected. Three user representatives have tested the questionnaire, and provided useful feedback resulting in minor revisions. Procedure. The study participants will fill in the questionnaire on the first and last course sessions. For the 6 and 15 months' follow-up, the participants will receive a SMS with a link to a common web page where the questionnaires may be completed. Digital data collection makes it easier to complete the questionnaires and ease the computing processes. The project will use external data management services that will program and test the digitalisation of the questionnaire. The data will be transferred into data files ready for use by the PhD candidate. Price estimates have been provided by suppliers of such services, and services will be acquired in line with public procurement policies. The PhD candidate will be in regular contact with the data management company and with HLC and NAV course leaders via email and telephone, ensuring timing of the SMSes to the measurement times. The PhD candidate will introduce the course leaders to the study during their two-day course leader training in 2020.

Data analysis. The effect analysis of the primary outcome will involve a comparison of self-reported wellbeing at course start and course end, using a two-way repeated (mixed) measures ANOVA. Additionally, longitudinal analyses will be conducted by fitting linear mixed (multilevel) models to data from all five time points. Mixed modelling is flexible and can handle non-balanced data with missing entries and repeated observations. The models allow the investigators to examine the effectiveness of the intervention and test hypotheses about group and individual trajectories in wellbeing, while controlling for both time variant and invariant covariates. Follow-up analyses will be conducted using various time-to-event approaches. Analyses will be performed in SPSS 25.0 (SPSS I, 2017) and R 3.5.3 (R Core Team 2019). Sample size and power. Simulations were performed in R 3.5.3 to assess power to detect an increase in wellbeing of 4.3 units from a baseline score of 12.5, the magnitude found in the pilot study, for each of the two subsamples (n=600 and n= 120) in both intervention and control groups, (sd=5, rho=0.5). Power to detect an interaction effect in mixed ANOVA (two tailed test, α=0.05) was found to be 1.0 (HLCs) and 1.0 (NAV), which is adequate, also allowing for dropout of 17 %. Although dropout is expected to increase for the later measurements, the multilevel analysis ensures utilisation of all available data. Power is higher in the linear mixed models, with data from additional three time points included for each participant.

The dissemination plan.

The dissemination plan will be the key tool to make the project findings available and relevant to the main stakeholders (users and staff), private, ideal and governmental users, the scientific community, and the media. The NCMH, core scientists and user groups will be actively involved in dissemination of all findings. Results from the project will be published in high quality open access international peer reviewed journals. Tentative titles of papers:

1. The 5 Ways to Wellbeing course: The effects on wellbeing, physical and mental health and mastery. A randomized controlled trial.
2. Reducing loneliness and improving social integration and social support: The long-term impact of the 5 Ways to Wellbeing course.
3. Effects of the 5 Ways to Wellbeing course on work participation in adults on sick leave and welfare benefits in The Norwegian Labour and Welfare Administration (NAV).

Additionally, results from the project will be published in condensed form accessible to both professionals and non-professionals by several means of dissemination. These include national conferences (e.g., HLC network conferences), Norwegian Institute of Public Health (NIPH) reports and newsletters, press releases for each scientific paper, and activity in social media.

ELIGIBILITY:
Inclusion Criteria:

* individuals with, or at high risk of disease, who need support in health behaviour change and in coping with health problems and chronic disease.
* individuals on sick leave, work assessment allowance (AAP) and disability pension

Exclusion Criteria:

* Severe mental illhealth
* impaired cognitive functioning

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Wellbeing | 15 months
  Diener's Flourishing scale, 2 items Scores is from 8 (lowest possible wellbeing) to 56 (highest possible wellbeing).
Wellbeing | 15 months
  Satisfaction With Life Scale (SWLS) scoring: 31 - 35 Extremely satisfied 26 - 30 Satisfied 21 - 25 Slightly satisfied 20 Neutral 15 - 19 Slightly dissatisfied 10 - 14 Dissatisfied 5 - 9 Extremely dissatisfied
Wellbeing | 15 months
  WHO-5

SECONDARY OUTCOMES:
Mental health | 15 months
  Patient Health Questionnaire-2, PHQ-2 Scores range from 0-6, the higher score the more depressed.
Mastery | 15 months
  Pearlin and Schooler's Mastery Scale Scores from 7-49, the higher score the higher mastery. Items 4 and 6 are reversed
Social life | 15 months
  Single question
Physical health | 15 months
  12-Item Short Form Survey (SF-12)/RAND-12 Scores: 12-47, where higher scores mean poorer health
Work participation | 15 months
  Single question
Health care usage | 15 months
  Single question

CONTACTS AND LOCATIONS:
Overall Officials: Anne Reneflot, PhD, Study Chair — Department Director
Locations (1):
- Norwegian Institute of Public Health, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No